CLINICAL TRIAL: NCT05650424
Title: The Effects of Infant Abdominal Massage on Postnatal Stress Level Among Chinese Parents in Hong Kong
Brief Title: Infant Abdominal Massage on Postnatal Stress Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lai Sze Ki, Principal Investigator, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HKUCTR-3008
Record Dates: First submitted 2022-12-01; First posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Parenting; Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wait-listed Control (Active Comparator): wait-listed control group will be put on wait list and receive abdominal massage class training on week 4 (posttest)
  Interventions: Other: Abdominal massage training
- Intervention (Receive abdominal massage training) (Experimental): Intervention group will receive abdominal massage training class and they will perform abdominal massage on their baby for 4 week. Parental stress level will be assessed on week 0 and week 4
  Interventions: Other: Abdominal massage training

INTERVENTIONS:
Other: Abdominal massage training — please refer to group description

SUMMARY:
The goal of this randomized control trial is to find out the effects of infant abdominal massage on postnatal stress level among Chinese parents in Hong Kong with babies under 1 year old. The main question[s] it aims to answer are:

* examine the effects of infant abdominal massage on postnatal stress level among Chinese parents in Hong Kong
* the relationship between the compliance of the intervention and the change of parental stress level Participants in intervention group will receive a abdominal massage training session and will perform on their baby. Parental stress level will be assess week 0 and four weeks .

If there is a comparison group: Researchers will compare wait-listed control group to see if there is any change on their parental stress level

DETAILED DESCRIPTION:
same as above

ELIGIBILITY:
Inclusion Criteria:

1. Parents aged 18 or above.
2. Parents with 0-1 year old full term babies without medical treatment of colic.
3. Able to communicate or read Chinese and have not tried applying infant massage on their babies.

Exclusion Criteria:

1. Parents with babies who had abdominal surgery.
2. Currently participating in any other massage related studies.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Parental stress level | week 4
  is parenting stress which was assessed by the parental stress scale of the Chinese version of the Parenting Stress Index (PSI-SF) (4th version) with 3 subscales: Difficult child (DC), Parental distress (PD) and Parent-child dysfunctional interaction (P-CDI)
  Total Score: 36-180 ( Higher score implies higher parental stress level)

SECONDARY OUTCOMES:
Difficult child | week 4
  Difficult child (DC) which is one of the subscales of PSI-SF
  Subscale score: 12-60 (Higher score mean a worse outcome)
Parental distress & Parent-child dysfunctional interaction | week 4
  Parental distress (PD) and Parent-child dysfunctional interaction (P-CDI) which are the other two subscales of PSI-SF
  Each Subscale score: 12-60 (Higher score mean a worse outcome)
Difference in parental stress with the presence of partner participation | week 4
  Difference in total parental stress level (PSI-SF) with the presence of partner participation to join the massage training class
Correlation between parental stress and self-reported compliance of the intervention | week 4
  Correlation between parental stress and self-reported compliance of the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lai VSK, Fong DYT. The effects of infant abdominal massage on the parental stress level among Chinese parents in Hong Kong - A mixed clustered RCT. BMC Complement Med Ther. 2024 Sep 28;24(1):342. doi: 10.1186/s12906-024-04636-6. PMID 39342220